CLINICAL TRIAL: NCT04334590
Title: Virtual Surgical Planning for the Fabrication of Sequential Naso-Alveolar Molding Appliances in the Treatment of Cleft Lip/Nose Deformities
Brief Title: Fabrication of Sequential Naso-Alveolar Molding Appliances in the Treatment of Cleft Lip/Nose Deformities
Status: Withdrawn | Type: Observational
Why Stopped: no enrollment
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00176186
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Cleft Lip; Congenital Nose Malformation; Deformity; Nose Deformities, Acquired
Keywords: Cleft Lip
MeSH Terms: conditions — Cleft Lip; Congenital Abnormalities; Nose Deformities, Acquired

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cleft Lip/Nose Repair without PSIO: Participants who will undergo cleft lip/nose repair prior to addition of PSIO as part of standard of care in Hopkins.
  Interventions: Procedure: Cleft Lip/Nose Repair without PSIO
- Presurgical Infant Orthopedic Therapy: Participants who will undergo cleft lip/nose repair after addition of PSIO as part of standard of care in Hopkins.
  Interventions: Procedure: Presurgical Infant Orthopedic Therapy

INTERVENTIONS:
Procedure: Cleft Lip/Nose Repair without PSIO — Standard of care surgical repair of cleft lip/nose without PSIO.
  Groups: Cleft Lip/Nose Repair without PSIO
Procedure: Presurgical Infant Orthopedic Therapy — Standard of care surgical repair of cleft lip/nose with PSIO.
  Groups: Presurgical Infant Orthopedic Therapy

SUMMARY:
There is a robust body of research suggesting that the use of pre-surgical orthopedic devices prior to definitive cleft lip/nose repair results in significant improvement of facial aesthetics with long term follow up. However, in recent surveys of the cleft centers in the US, only 30% of cleft centers offer PSIOs, and only 13% routinely report its use. Accordingly, thirty percent of centers utilize a two-stage cleft lip/nose repair in the centers' algorithm (1st: lip adhesion; 2nd: final lip repair). The major drawback to a two-stage cleft procedure is the administration of two general anesthetics to an infant before the age of one year. There is a growing amount of evidence that multiple anesthetic experiences before a certain age could affect brain development.

It is difficult to make inferences as to why clinicians are not utilizing surgical aids to decrease the size of the cleft width, but even when PSIO is offered, caregivers experience additional, potentially prohibitive challenges. In one study, caregivers traveled an average of 70 miles to visit the nearest cleft center offering pre-surgical orthopedic devices. As these devices are created by hand every 1-2 weeks after seeing the child in clinic, parents are required to travel to clinic multiple times per month. Not surprisingly, infants who were first-born and those who did not have other siblings were more likely to receive pre-surgical orthopedic treatment than infants who were residing with other siblings.

Given the benefits of PSIOs and the barriers both to healthcare systems and patients' families associated with PSIOs in its current form, a new form of pre-surgical clinical management is needed.

Objectives:

1. Evaluate JHH's current clinical performance in addressing unilateral cleft lip and nasal deformity.
2. Elucidate the difference in preoperative cleft size and in surgical management/outcomes for patients who received PSIOs through 3D-printed devices.
3. Using the above maxillofacial growth data with and without PSIOs, the investigators aim to create an algorithm to predict maxillofacial growth for each individual patient to design pre-sequenced custom PSIO devices.

DETAILED DESCRIPTION:
Approximately 7000 babies are born with a cleft lip and/or cleft palate in the United States per year. Globally, this defect is staggeringly common, with 100,000 new cases per year. This defect is due to a failure of normal fusion between facial structures, causing a full thickness gap of the upper lip involving skin, muscle, and other connective tissue. Due to aberrant insertion of the muscle underlying the lip as well as abnormal formation of deeper facial structures, the nose is also displaced inferiorly, laterally, and posteriorly. The wider the cleft, the more challenging the repair.

Current best practice in treating unilateral cleft lip and nose deformity involves presurgical infant orthopedics (PSIOs). PSIOs involves presurgically treating the deformity using custom orthodontics to gradually bring the two halves of the cleft together, reducing defect size and enabling complete repair with one surgery during early infancy. However, creation of these molds is time consuming and requires the expertise of a cleft orthodontist and weekly visits to the hospital for device advancement. As not all cleft centers have a specialized cleft orthodontist-including Johns Hopkins Hospital-many are unable to provide presurgical infant orthopedics. Weekly travel to cleft centers can also pose a significant temporal and financial burden to families, as the average patient is located over 60 miles from the nearest cleft center. In a recent survey of cleft centers in the United States, only 30% of these centers are able to provide presurgical orthopedic molding devices in treatment protocols. These centers therefore correct wide clefts with a staged, two-surgery approach. This approach is often less successful in both adequately aligning the gum and in repairing nasal defects, and usually requires intensive orthodontics and additional surgeries in adolescence. As the defect is not fully corrected in infancy, children are additionally subjected to the emotional and psychological difficulty and damage to self-esteem associated with the persistent defect.

With the advent of 3D printing technology, the investigators are now in the planning stages of implementing a new clinical protocol to bring PSIOs to Johns Hopkins Hospital (JHH). A cleft orthodontist at an equipped center will remotely design these orthodontic molds, which will then be 3D printed using dental acrylic (the same material currently used in hand-fabricated orthodontic models) and given to patients in the investigators' clinic. As planning these devices for 3D printing can be done remotely in a fraction of the time it would take to create each one by hand, this change in clinical practice will eliminate the need for an in-person specialized craniofacial orthodontist on faculty where one does not exist.

This research study seeks to elucidate both the investigators' current standard of cleft practice and the benefits the investigators hope to see after implementing this change in clinical practice. The investigators expect that although the investigators will initially create each new mold after a weekly hospital visit with in-person measurements, the investigators ultimately aim to develop an algorithm to predict early growth and development of the newborn's facial skeleton and soft tissue. This will allow the fabrication of sequential pre-surgical orthopedic molding devices based of the infant's predicted facial growth, which can be delivered en bloc to the infants home, thereby eliminating the need for frequent visits to geographically inconvenient centers. After 4-5 months of using these devices, the bony cleft gap will be closed, the nose straightened, and the child be ready for the definitive cleft lip and nose repair in a single surgery. These devices will not only physically close the gap of the cleft lip deformity, but will also close the gap in access to the necessary specialists for the ideal management of cleft deformities across the country. With this technology, any cleft center can offer naso-alveolar molding to every child born with cleft lip and palate in the country.

ELIGIBILITY:
Inclusion Criteria:

* All newborns either born in Johns Hopkins or presenting to clinic with a cleft lip between 0-1 months of life

Exclusion Criteria:

* Patients older than one month of age at presentation

Ages: 0 Months to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborns either born in Johns Hopkins or presenting to clinic with a cleft lip between 0-1 months of life.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of cleft patients with an alveolar cleft of <5 mm at time of the first surgery | At the time of first surgery (3 months)
  Percentage of cleft patients with an alveolar cleft of <5 mm at time of the first surgery will be assessed to determine the effect of 3D printed orthognathic pre-surgical molding devices on cleft care.
Cleft size at initial clinic presentation | At the time of initial clinic visit up to 1 hour
  Cleft size in millimeters (mm) at initial clinic presentation.
Size of cleft at pre- and post-operative clinic visit | At pre- and post-operative clinic visit, up to 4 months
  Size of cleft in millimeters at pre- and post-operative clinic visit

SECONDARY OUTCOMES:
Rate of change in cleft size | Weekly, up 8 weeks
  The rate of change in cleft size (mm/week).
Length of time to achieve a cleft <5 mm | Up to 4 months
  Length of time in days to achieve a cleft <5 mm.
Aesthetic outcome following cleft surgical repair as assessed by the surgeon | Post surgery, up to 4 months
  Aesthetic outcome following cleft surgical repair wiil be assessed by the surgeon using a clinical judgment.
Satisfaction with the 3-D printed pre-surgical orthopedic device as assessed by parents | Post surgery, up to 4 months
  Satisfaction with the 3-D printed pre-surgical orthopedic device will be assessed by a satisfaction questionnaire administered to parents.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Redett, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States